CLINICAL TRIAL: NCT06230991
Title: A Pilot Study of Efficacy and Safety of a Microbiome Immunity Formula (SIM05) in Adults With Atopic Eczema
Brief Title: A Pilot Study of Efficacy and Safety of SIM05 in Adults With Atopic Eczema
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AEZ-SIM05
Record Dates: First submitted 2023-10-30; First posted 2024-01-30 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Atopic Eczema
Keywords: Atopic Eczema; Gut Microbiota; Probiotics
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: All study subjects will receive the same study products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SIM05 (Experimental): One sachet twice daily for 16 weeks
  Interventions: Dietary Supplement: SIM05

INTERVENTIONS:
Dietary Supplement: SIM05 — SIM05 contains a blend of food-grade Bifidobacterium and Lactobacillus strains plus prebiotics
  Other Names: G-NiiB immunity formula

SUMMARY:
Atopic eczema causes significant disease burdens worldwide. Some studies reported gastrointestinal symptoms in eczema patients which could be related to gut microbiota change. A unique gastrointestinal microflora pattern has also been observed in atopic dermatitis patients when compared with healthy controls. To date, no adult formula is specific for alleviating atopic eczema-related symptoms (especially through change of gut microbiota) for adults. The investigators hypothesize that the gut microbiota of adults with atopic eczema can be modulated to decrease the severity of atopic eczema-related symptoms. A pilot study is proposed to assess the effect and safety of SIM05 on atopic eczema severity and gut microbiome of adults with atopic eczema.

DETAILED DESCRIPTION:
The major atopic disorders, atopic eczema, allergic rhinitis and asthma, cause significant disease burdens worldwide.

Apart from cutaneous symptoms such as dryness and itchiness in eczema patients [4], studies also reported gastrointestinal symptoms which could be related to gut microbiota change. Unique gastrointestinal microflora pattern has also been observed in atopic dermatitis patients when compared with healthy controls: decreased Bifidobacterium and Enterococci, especially Bifidobacterium bifidum and Bifidobacterium longum, and increased Faecalibacterium have been observed. Therefore, gastrointestinal microflora can serve as the disease indicator of atopic eczema. Emerging evidence also suggests that gut microbiota modulation can largely affect host immune functions in adults.

To date, no adult formula is specific for alleviating atopic eczema-related symptoms (especially through change of gut microbiota) for adults. SIM05 contains a blend of naturally occurring three food-grade probiotics strains and three prebiotics. The three probiotics belong to food-grade Bifidobacterium and Lactobacillus, which is an important group of probiotic cultures commonly used in food products. Moreover, research showed that Lactobacillus and Bifidobacteria could prevent atopic sensitisation to common food allergens and thus reducing the incidence of atopic eczema.

The investigators hypothesize that the gut microbiota of adult with atopic eczema can be modulated to decrease the severity of atopic eczema related symptoms. A pilot study of 30 adults with atopic eczema who will receive SIM05 for 16 weeks is proposed to assess the effect and safety of SIM05 on atopic eczema severity and gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or older physician-diagnosed atopic eczema;
* Agree to sign the informed consent form

Exclusion Criteria:

* Adults with other documented chronic and clinically significant dermatologic diseases that may interfere with the evaluation of cutaneous signs and symptoms. Common conditions such as acne are permissible.
* Adults with atopic eczema who have taken antibiotics within one months prior to recruitment.
* Adults with atopic eczema who require systemic immunosuppressive treatments (e.g. azathioprine, methotrexate, mycophenolate mofetil, cyclosporine, biologics) within three months prior to recruitment, or who are taking systemic steroids within one month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Change in Eczema Area and Severity Index (EASI) across 16 weeks. | 16 weeks
  The change of score in Eczema Area and Severity Index. A score of 0 indicates clear or no eczema, 0.1 to 1.0 indicates almost clear, 1.1 to 7 indicates mild disease, 7.1 to 21 indicates moderate disease, 21.1 to 50 indicates severe disease, and greater than 51 indicates very severe disease.

SECONDARY OUTCOMES:
Percentage of subjects achieving 50% and 75% reduction in EASI (EASI-50, EASI-75). | 16 weeks
  The percentage reduction in EASI score
Change in pruritus numerical rating scales (pruritus-NRS) across 16 weeks. | 16 weeks
  The change of quality of life measuring in pruritus-NRS. On a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable".
Changes in faecal microbial profiling across 16 weeks. | 16 weeks
  The changes of profile in faecal microbial
Adverse events reported during the study period. | 16 weeks
  The adverse events reported throughout the study
Change in Dermatology life quality index (DLQI) across 16 weeks. | 16 weeks
  The change of quality of life measuring in DLQI scales. The scoring of each question is 'very much = 3'; 'quite a lot = 2'; 'only a little = 1' and 'not at all = 0'. The meaning of scores: 0-1 = no effect on life; 2-6 = small effect; 7-12 = moderate effect; 13-18 = very large effect and 19-30 = extremely large effect.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Ching, PhD, Study Director — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng NS, Chau JPC, Lo SHS, Choi KC, Hon KLE, Lam PH, Leung TF. Effects of a self-efficacy theory-based parental education program on eczema control and parental outcomes. Pediatr Allergy Immunol. 2021 Apr;32(3):535-543. doi: 10.1111/pai.13421. Epub 2020 Dec 4. PMID 33274772
- [Background] Makrgeorgou A, Leonardi-Bee J, Bath-Hextall FJ, Murrell DF, Tang ML, Roberts A, Boyle RJ. Probiotics for treating eczema. Cochrane Database Syst Rev. 2018 Nov 21;11(11):CD006135. doi: 10.1002/14651858.CD006135.pub3. PMID 30480774
- [Background] Chan CX, Zug KA. Diagnosis and Management of Dermatitis, Including Atopic, Contact, and Hand Eczemas. Med Clin North Am. 2021 Jul;105(4):611-626. doi: 10.1016/j.mcna.2021.04.003. PMID 34059241
- [Background] Kimata H. Modulation of fecal polyamines by viewing humorous films in patients with atopic dermatitis. Eur J Gastroenterol Hepatol. 2010 Jun;22(6):724-8. doi: 10.1097/MEG.0b013e32832e09f1. PMID 19543102
- [Background] Silverberg JI, Hanifin JM. Adult eczema prevalence and associations with asthma and other health and demographic factors: a US population-based study. J Allergy Clin Immunol. 2013 Nov;132(5):1132-8. doi: 10.1016/j.jaci.2013.08.031. Epub 2013 Oct 4. PMID 24094544
- [Background] Watanabe S, Narisawa Y, Arase S, Okamatsu H, Ikenaga T, Tajiri Y, Kumemura M. Differences in fecal microflora between patients with atopic dermatitis and healthy control subjects. J Allergy Clin Immunol. 2003 Mar;111(3):587-91. doi: 10.1067/mai.2003.105. PMID 12642841
- [Background] Burr S. Assessment and management of eczema in adults in the community setting. Br J Community Nurs. 2019 Mar 2;24(3):110-115. doi: 10.12968/bjcn.2019.24.3.110. No abstract available. PMID 30817210
- [Background] Song H, Yoo Y, Hwang J, Na YC, Kim HS. Faecalibacterium prausnitzii subspecies-level dysbiosis in the human gut microbiome underlying atopic dermatitis. J Allergy Clin Immunol. 2016 Mar;137(3):852-60. doi: 10.1016/j.jaci.2015.08.021. Epub 2015 Oct 1. PMID 26431583
- [Background] Quince C, Walker AW, Simpson JT, Loman NJ, Segata N. Shotgun metagenomics, from sampling to analysis. Nat Biotechnol. 2017 Sep 12;35(9):833-844. doi: 10.1038/nbt.3935. PMID 28898207
- [Background] Pugh JN, Sparks AS, Doran DA, Fleming SC, Langan-Evans C, Kirk B, Fearn R, Morton JP, Close GL. Four weeks of probiotic supplementation reduces GI symptoms during a marathon race. Eur J Appl Physiol. 2019 Jul;119(7):1491-1501. doi: 10.1007/s00421-019-04136-3. Epub 2019 Apr 13. PMID 30982100
- [Background] Prasanna PHP, Grandison AS, Charalampopoulos D. Bifidobacteria in milk products: An overview of physiological and biochemical properties, exopolysaccharide production, selection criteria of milk products and health benefits. Food Res Int 2014;55:247-62.
- [Background] Hanifin JM, Baghoomian W, Grinich E, Leshem YA, Jacobson M, Simpson EL. The Eczema Area and Severity Index-A Practical Guide. Dermatitis. 2022 May-Jun 01;33(3):187-192. doi: 10.1097/DER.0000000000000895. PMID 35594457
- [Background] Simpson EL, Bieber T, Guttman-Yassky E, Beck LA, Blauvelt A, Cork MJ, Silverberg JI, Deleuran M, Kataoka Y, Lacour JP, Kingo K, Worm M, Poulin Y, Wollenberg A, Soo Y, Graham NM, Pirozzi G, Akinlade B, Staudinger H, Mastey V, Eckert L, Gadkari A, Stahl N, Yancopoulos GD, Ardeleanu M; SOLO 1 and SOLO 2 Investigators. Two Phase 3 Trials of Dupilumab versus Placebo in Atopic Dermatitis. N Engl J Med. 2016 Dec 15;375(24):2335-2348. doi: 10.1056/NEJMoa1610020. Epub 2016 Sep 30. PMID 27690741
- [Background] Guttman-Yassky E, Teixeira HD, Simpson EL, Papp KA, Pangan AL, Blauvelt A, Thaci D, Chu CY, Hong HC, Katoh N, Paller AS, Calimlim B, Gu Y, Hu X, Liu M, Yang Y, Liu J, Tenorio AR, Chu AD, Irvine AD. Once-daily upadacitinib versus placebo in adolescents and adults with moderate-to-severe atopic dermatitis (Measure Up 1 and Measure Up 2): results from two replicate double-blind, randomised controlled phase 3 trials. Lancet. 2021 Jun 5;397(10290):2151-2168. doi: 10.1016/S0140-6736(21)00588-2. Epub 2021 May 21. PMID 34023008
- [Background] Heinl D, Prinsen CA, Deckert S, Chalmers JR, Drucker AM, Ofenloch R, Humphreys R, Sach T, Chamlin SL, Schmitt J, Apfelbacher C. Measurement properties of adult quality-of-life measurement instruments for eczema: a systematic review. Allergy. 2016 Mar;71(3):358-70. doi: 10.1111/all.12806. Epub 2015 Dec 16. PMID 26564008
- [Background] Yosipovitch G, Reaney M, Mastey V, Eckert L, Abbe A, Nelson L, Clark M, Williams N, Chen Z, Ardeleanu M, Akinlade B, Graham NMH, Pirozzi G, Staudinger H, Plaum S, Radin A, Gadkari A. Peak Pruritus Numerical Rating Scale: psychometric validation and responder definition for assessing itch in moderate-to-severe atopic dermatitis. Br J Dermatol. 2019 Oct;181(4):761-769. doi: 10.1111/bjd.17744. Epub 2019 May 1. PMID 30729499
- [Background] Silverberg NB. Typical and atypical clinical appearance of atopic dermatitis. Clin Dermatol. 2017 Jul-Aug;35(4):354-359. doi: 10.1016/j.clindermatol.2017.03.007. Epub 2017 Mar 24. PMID 28709565